CLINICAL TRIAL: NCT02931357
Title: A Randomized, Open, Parallel-group Multicenter Study of Efficacy and Tolerability of a New Medical Device in Gel Formulation (Hyaluronic Acid 0.54%) Versus Calgel® for the Topical Treatment of Teething in Infants
Brief Title: Study of a New Medical Device in Gel Formulation Versus Calgel® for the Topical Treatment of Teething in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ricerfarma S.r.l (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other); Latis S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GENG10-12
Record Dates: First submitted 2016-09-29; First posted 2016-10-13 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Pain Teeth
Keywords: Treatment of teething in infants
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic Acid 0.54% (Experimental): Administration: application of the gel on the gingival tissue, massage it in gently, five to six times a day.
  Interventions: Device: Hyaluronic Acid 0.54%
- Calgel® (Active Comparator): Administration: application of the gel on the gingival tissue, massage it in gently, three/four times a day (away from meals). In any case the interval between gel applications must be at least 3 hours.
  Interventions: Drug: Calgel®

INTERVENTIONS:
Device: Hyaluronic Acid 0.54% — Administration: application of the gel on the gingival tissue, massage it in gently, five to six times a day
  Other Names: Hyaluronic Acid gel 0.54%.
  Arms: Hyaluronic Acid 0.54%
Drug: Calgel® — Administration: application of the gel on the gingival tissue, massage it in gently, three/four times a day (away from meals). In any case the interval between gel applications must be at least 3 hours.
  Other Names: Lidocaine 0.33% and Cetylpyridinium Chloride 0.10%
  Arms: Calgel®

SUMMARY:
This is a randomized, open label, parallel-groups, multicenter study. The study will be conducted in three clinical sites. Test Medical Device: 0.54% Hyaluronic Acid rose honey flavour gel medical device class IIa.

DETAILED DESCRIPTION:
Due to the potentially serious toxicity that can result from the use of topical anesthetics to relieving the symptoms associated with gingival inflammatory conditions or gums trauma in infant, recently, products containing Hyaluronic Acid have been marketed in Europe. In particular, Ricerfarma is developing several high molecular weight Hyaluronic Acid medical devices characterized by the absence of preservatives, alcohol and dyes; therefore, the administration of these products in infants is safe and can help creating a natural protective layer on the gingival tissue. In previous clinical trials with these high molecular weight Hyaluronic Acid medical devices it was noted a periodontal tissue/fluid balance with accelerated healing and repair properties that could be of interest either for accelerating the wound healing process or for treating the complex physical symptoms (i.e. soreness and swelling of gums, crying, sleeplessness) related to the teething in infants. These data were confirmed by a recent pilot study on 18 infants suffering by teething where the two formulation of the tested high molecular weight Hyaluronic Acid medical device evidenced, at the end of treatment period, for pain, swelling, gingival rush, hyper-salivation and redness a statistically significant reduction from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infants aged between 6 and 36 months.
2. Teething diagnosed by the presence of at least 3 of the following clinical symptoms:

   pain, swelling, gingival rush, hyper-salivation, redness, abnormal teeth depth.
3. At the moment of inclusion no subcutaneous mucosal laceration must be yet appeared.
4. Informed consent form signed by parents or legal representative.
5. Infants and parents who are in a general position to follow all study requirements

Exclusion Criteria:

1. Infants in hospitalization and/or immobilization and/or confinement to bed.
2. Infants with known history of severe renal insufficiency and/or known history of severe cardiac dysfunction and/or liver problems
3. Use of topical Lidocaine and/or topical Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) within one day before inclusion.
4. Use of systemic NSAIDs within 3 days before inclusion and/or use of systemic anesthetics within 10 days before.
5. Concomitant use during the period of study of NSAIDs and/or any anesthetics (obviously Calgel® is allowed in patients randomized in group B, only)
6. Subjects with known history of allergic or adverse reactions to avian proteins or to HA and to any ingredient of the Medical Device and/or of the comparator on study.
7. Infants whose parents suffer from any form of psychiatric disorder or other condition which, in the opinion of the Investigator, might invalidate the required prescription and/or observation or complicate communication with the subject.
8. Infants simultaneously participating or having participated in the last month before Visit 1 in another clinical trial.
9. Infants already treated under this protocol.

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Teething pain | day 0, 3 and 7
  scored according to intensity with the following Verbal Rating Scale: Absent = 0, Moderate = 1, Intense = 2

SECONDARY OUTCOMES:
day pain | day 0, 3 and 7
  scored according to intensity with the following Verbal Rating Scale: Absent = 0, Moderate = 1, Intense = 2
gingival rush | day 0, 3 and 7
  scored according to intensity with the following Verbal Rating Scale: Absent = 0, Moderate = 1, Intense = 2
hyper-salivation | day 0, 3 and 7
  scored according to intensity with the following Verbal Rating Scale: Absent = 0, Moderate = 1, Intense = 2
redness | day 0, 3 and 7
  scored according to intensity with the following Verbal Rating Scale: Absent = 0, Moderate = 1, Intense = 2
swelling | day 0, 3 and 7
  scored according to intensity with the following Verbal Rating Scale: Absent = 0, Moderate = 1, Intense = 2

CONTACTS AND LOCATIONS:
Overall Officials: Serban Rosu, MD, Principal Investigator — Societatea Civile Medicala Dr.Rosu
Locations (1):
- Opera Contract Research Organization SRL, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pytlik W. [Symptoms of the failure of the biological mechanism of teething. Symptomatology of the primary teeth's reinclusion]. Czas Stomatol. 1989 Jan;42(1):29-34. Polish. PMID 2640634
- [Background] McIntyre GT, McIntyre GM. Teething troubles? Br Dent J. 2002 Mar 9;192(5):251-5. doi: 10.1038/sj.bdj.4801349. PMID 11924952
- [Background] Owais AI, Zawaideh F, Al-Batayneh OB. Challenging parents' myths regarding their children's teething. Int J Dent Hyg. 2010 Feb;8(1):28-34. doi: 10.1111/j.1601-5037.2009.00412.x. PMID 20096079
- [Background] Curtis LA, Dolan TS, Seibert HE. Are one or two dangerous? Lidocaine and topical anesthetic exposures in children. J Emerg Med. 2009 Jul;37(1):32-9. doi: 10.1016/j.jemermed.2007.11.005. Epub 2008 Feb 14. PMID 18280086
- [Background] Weigel PH, Fuller GM, LeBoeuf RD. A model for the role of hyaluronic acid and fibrin in the early events during the inflammatory response and wound healing. J Theor Biol. 1986 Mar 21;119(2):219-34. doi: 10.1016/s0022-5193(86)80076-5. PMID 3736072
- [Background] Bartold PM. The effect of interleukin-1 beta on hyaluronic acid synthesized by adult human gingival fibroblasts in vitro. J Periodontal Res. 1988 Mar;23(2):139-47. doi: 10.1111/j.1600-0765.1988.tb01347.x. No abstract available. PMID 2967366
- [Background] Oksala O, Salo T, Tammi R, Hakkinen L, Jalkanen M, Inki P, Larjava H. Expression of proteoglycans and hyaluronan during wound healing. J Histochem Cytochem. 1995 Feb;43(2):125-35. doi: 10.1177/43.2.7529785.
- [Background] Irwin CR, Schor SL, Ferguson MW. Effects of cytokines on gingival fibroblasts in vitro are modulated by the extracellular matrix. J Periodontal Res. 1994 Sep;29(5):309-17. doi: 10.1111/j.1600-0765.1994.tb01227.x. PMID 7799210
- [Background] Pistorius A, Martin M, Willershausen B, Rockmann P. The clinical application of hyaluronic acid in gingivitis therapy. Quintessence Int. 2005 Jul-Aug;36(7-8):531-8. PMID 15999421
- [Background] Brandt FS, Cazzaniga A. Hyaluronic acid gel fillers in the management of facial aging. Clin Interv Aging. 2008;3(1):153-9. doi: 10.2147/cia.s2135. PMID 18488885
- [Background] Dagenais S. Intra-articular hyaluronic acid (viscosupplementation) for knee osteoarthritis. Issues Emerg Health Technol. 2006 Nov;(94):1-4. PMID 17096501
- [Background] Fernandez Lopez JC, Ruano-Ravina A. Efficacy and safety of intraarticular hyaluronic acid in the treatment of hip osteoarthritis: a systematic review. Osteoarthritis Cartilage. 2006 Dec;14(12):1306-11. doi: 10.1016/j.joca.2006.08.003. Epub 2006 Sep 18. PMID 16979914
- [Background] Iavazzo C, Athanasiou S, Pitsouni E, Falagas ME. Hyaluronic acid: an effective alternative treatment of interstitial cystitis, recurrent urinary tract infections, and hemorrhagic cystitis? Eur Urol. 2007 Jun;51(6):1534-40; discussion 1540-1. doi: 10.1016/j.eururo.2007.03.020. Epub 2007 Mar 20. PMID 17383810
- [Background] Liguori V, Guillemin C, Pesce GF, Mirimanoff RO, Bernier J. Double-blind, randomized clinical study comparing hyaluronic acid cream to placebo in patients treated with radiotherapy. Radiother Oncol. 1997 Feb;42(2):155-61. doi: 10.1016/s0167-8140(96)01882-8. PMID 9106924
- [Background] Igic M, Mihailovic D, Kesic L, Apostolovic M, Kostadinovic L, Janjic OT, Milasin J. [Efficacy of hyaluronic acid in the treatment of chronic gingivitis in children]. Vojnosanit Pregl. 2011 Dec;68(12):1021-5. doi: 10.2298/vsp1112021i. Serbian. PMID 22352262
- [Background] Mesa FL, Aneiros J, Cabrera A, Bravo M, Caballero T, Revelles F, del Moral RG, O'Valle F. Antiproliferative effect of topic hyaluronic acid gel. Study in gingival biopsies of patients with periodontal disease. Histol Histopathol. 2002;17(3):747-53. doi: 10.14670/HH-17.747. PMID 12168783
- [Background] Moseley R, Waddington RJ, Embery G. Hyaluronan and its potential role in periodontal healing. Dent Update. 2002 Apr;29(3):144-8. doi: 10.12968/denu.2002.29.3.144. PMID 11989392
- [Background] Nolan A, Baillie C, Badminton J, Rudralingham M, Seymour RA. The efficacy of topical hyaluronic acid in the management of recurrent aphthous ulceration. J Oral Pathol Med. 2006 Sep;35(8):461-5. doi: 10.1111/j.1600-0714.2006.00433.x. PMID 16918596
- [Background] Nolan A, Badminton J, Maguire J, Seymour RA. The efficacy of topical hyaluronic acid in the management of oral lichen planus. J Oral Pathol Med. 2009 Mar;38(3):299-303. doi: 10.1111/j.1600-0714.2008.00739.x. PMID 19267842